CLINICAL TRIAL: NCT05615922
Title: Remotely Supervised Transcranial Direct Current Stimulation (tDCS) for Primary Progressive Aphasia (PPA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-01155
Record Dates: First submitted 2022-11-03; First posted 2022-11-14 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Primary Progressive Aphasia
Keywords: Transcranial Direct Current Stimulation (tDCS)
MeSH Terms: conditions — Aphasia, Primary Progressive | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Remotely Supervised tDCS and Word-Naming Practice (Experimental): At each session, the tDCS device will deliver 2.0 mA electric current for 30 minutes over the left frontotemporal lobe with focus on the inferior frontal gyrus (IFG). Participants will receive 20 intervention sessions over the course of the interventional period (4 weeks) on weekdays (Monday-Friday). During the stimulation period, participants will engage in a picture-naming exercise as guided by the study tDCS clinicians.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS); Behavioral: Word-Naming Activity

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (tDCS) — tDCS is noninvasive brain stimulation device that modulates brain activity by delivering a low-intensity electrical current (2.0 mA) through scalp sponge electrodes. The device is preprogrammed to ramp up to 2.0 mA (for 30 seconds), provide constant current throughout session (29 minutes), and then ramp down (for 30 seconds) at the end.
  Other Names: Soterix Medical mini-CT Model 1601-LTE Stimulator
Behavioral: Word-Naming Activity — During each tDCS session, the tDCS clinician will guide the participant in a word-naming exercise. Participants will be presented with photos of target items and prompted to verbally produce the names of the pictures.

SUMMARY:
The purpose of this study is to establish the feasibility of a program of remotely supervised transcranial direct current stimulation (RS-tDCS) paired with language skills practice for people living with the semantic or logopenic variants of primary progressive aphasia (PPA). There are currently no established standard-of-care treatments for PPA. This study will evaluate whether RS-tDCS combined with language skills practice is a feasible study design for individuals with PPA.

ELIGIBILITY:
Inclusion Criteria:

1. Primary progressive aphasia diagnosis (logopenic or semantic variant)
2. Peabody Picture Vocabulary Test (PPVT) score < -1.0 SD, serving as a literacy proxy for premorbid cognitive ability and ensuring English language fluency sufficient for participation in the study procedures.
3. WAIS-IV Matrix Reasoning T score < 20, serving as an index of current general cognitive functioning to exclude those with severe cognitive impairment
4. Stable and continuous access to internet service, email (WiFi "hotspot" to be provided if needed)
5. Fluent in English language (due to outcomes validated in English versions only)

Exclusion Criteria:

1. Disorder other than PPA known to cause language dysfunction
2. Diagnosis of nonfluent/agrammatic subtype of primary progressive aphasia
3. History of traumatic brain injury
4. Uncontrolled seizure disorder and/or recent (<5 years) history of seizure
5. Metal implants in the head or neck
6. Any skin disorder or skin sensitive area near stimulation locations
7. Pregnant or breastfeeding

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-12-24 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2023-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leigh Charvet, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: [leigh.charvet@nyulangone.org]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to leigh.charvet@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Remotely Supervised tDCS and Word-Naming Practice
Started | 11
Completed | 10
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Remotely Supervised tDCS and Word-Naming Practice
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Complete 16 Out of 20 Study Visits
Description: Measure of feasibility.
Time Frame: Week 4
Measure: Number; unit: percentage of participants
Arm/Group | Remotely Supervised tDCS and Word-Naming Practice
Number analyzed (Participants) | 10
percentage of participants | 100

2. Secondary Outcome: Number of Trained Language Probes at Treatment End
Description: At baseline participants were shown photos of common items and assessed for spontaneous naming of each item. Thirty items were then selected for participants to be trained on, and 30 items served as the control word naming list. At study end, participants were assessed on their ability to spontaneously name the target words without the need for cueing.
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: Number of Trained Language Probes
Arm/Group | Remotely Supervised tDCS and Word-Naming Practice
Number analyzed (Participants) | 10
Number of Trained Language Probes | 25.1 (4.33)

3. Secondary Outcome: Number of Untrained Language Probes at Treatment End
Description: as for outcome 2
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: Number of Untrained Language Probes
Arm/Group | Remotely Supervised tDCS and Word-Naming Practice
Number analyzed (Participants) | 10
Number of Untrained Language Probes | 20.2 (7.07)

4. Secondary Outcome: Change in Aphasia Communication Outcome Measure (ACOM) Score
Description: Measurement of patient-reported communicative functioning in aphasia. Scores are presented as T-Scores that range from 0 to 100 with 50 representing the mean, with a standard deviation of ±10 indicating greater/less than average; higher T-scores indicate greater functional communication skills.
Time Frame: Baseline, Month 6
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Remotely Supervised tDCS and Word-Naming Practice
Number analyzed (Participants) | 10
T-score | 0.74 (0.77)

5. Secondary Outcome: Change in Stroke and Aphasia Quality of Life-39 Item (SAQOL-39) Score
Description: 39-item assessment of quality of life among individuals with aphasia. Items are ranked on a Likert scale ranging from 1 (Couldn't do it at all) to 5 (No trouble at all). The total score is the average score of all items and ranges from 1 to 5; higher scores indicate greater quality of life.
Time Frame: Baseline, Month 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Remotely Supervised tDCS and Word-Naming Practice
Number analyzed (Participants) | 10
score on a scale | -0.07 (0.2)

6. Secondary Outcome: Change in Patient-Reported Outcomes Measurement Information System (PROMIS) - Social Roles and Activities Score
Description: 35-item measurement of the perceived ability to perform one's usual social roles and activities. Each item is rated on a Likert scale ranging from 5 (never) to 1 (always). The raw score is the sum of responses and is converted to a T-score that has a population mean score of 50 with a standard deviation of 10; higher scores indicate greater ability to perform social roles and activities.
Time Frame: Baseline, Month 6
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Remotely Supervised tDCS and Word-Naming Practice
Number analyzed (Participants) | 10
T-score | -1.2 (3.48)

7. Secondary Outcome: Change in Patient-Reported Outcomes Measurement Information System (PROMIS) - Global Health Score
Description: 10-item measurement of symptoms, functioning, and healthcare-related quality of life. The raw score is the sum of responses and is converted to a T-score that has a population mean score of 50 with a standard deviation of 10; higher scores indicate better QOL.
Time Frame: Baseline, Month 6
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Remotely Supervised tDCS and Word-Naming Practice
Number analyzed (Participants) | 10
T-score | 0.87 (0.89)

8. Secondary Outcome: Change in Quick Aphasia Battery (QAB) Score
Description: Assessment of language function. Includes eight subtests, each of which comprise sets of items that probe different language domains, vary in difficulty, and are scored with a graded system to maximize the informativeness of each item. The total scores range from 0 to 10, where:
  * 0.00-4.99 = Severe Aphasia
  * 5.00-7.49 = Moderate Aphasia
  * 7.50-8.89 = Mild Aphasia
  * 8.90-10.00 = No Aphasia
Time Frame: Baseline, Month 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Remotely Supervised tDCS and Word-Naming Practice
Number analyzed (Participants) | 10
score on a scale | 0.14 (0.31)

9. Secondary Outcome: Change in Boston Naming Test (BNT)-Short Form Score
Description: Measures confrontational word retrieval in individuals with aphasia or other language disturbance. Consists of 15 line-drawn pictures presented in order of difficulty from "easiest" (e.g., "house") to "most difficult" (e.g., "palette"). Participants have 20 seconds to name each item correctly with a cueing hierarchy. The total score is the sum of correct responses and ranges from 0 to 15; higher scores indicate greater confrontational word retrieval abilities.
Time Frame: Baseline, Month 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Remotely Supervised tDCS and Word-Naming Practice
Number analyzed (Participants) | 10
score on a scale | 1.6 (0.37)

10. Secondary Outcome: Change in Controlled Oral Word Association Test (COWAT) Score
Description: The COWAT is verbal fluency test that measures spontaneous production of words belonging to the same category or beginning with some designated letter. The participants' task is to produce as many words as possible that begin with the given letter (F, A, or S) within a 1-minute time period. The total score is the total number of acceptable words produced for all three letters. The lowest possible score is zero, meaning no words could be produced. There is no limit to the higher end of the scale given that participants can produce as many words as possible for each of the three letters. Higher scores indicate greater word retrieval and better cognitive function.
Time Frame: Baseline, Month 6
Measure: Mean (Standard Deviation); unit: Correct words
Arm/Group | Remotely Supervised tDCS and Word-Naming Practice
Number analyzed (Participants) | 10
Correct words | 1.4 (2.23)

ADVERSE EVENTS:
Time Frame: All reportable events will be recorded with start dates occurring any time after informed consent is obtained until 7 months (4 weeks of intervention + follow-up at 6 months) (for non-serious AEs) or 30 days (for SAEs) after the last day of study participation
Description: Systematic, via check in with participant in advance of each treatment session with capture of any spontaneous reports
Arm/Group | Remotely Supervised tDCS and Word-Naming Practice
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-27): https://cdn.clinicaltrials.gov/large-docs/22/NCT05615922/Prot_SAP_000.pdf